CLINICAL TRIAL: NCT03850860
Title: Comparison of the Tolerance of Vancomycin in Combination With Piperacillin/Tazobactam or Cefepim as Empirical Antimicrobial Therapy of Prosthetic Joint Infection
Brief Title: Comparison of Two Empirical Antimicrobial Therapies of Prosthetic Joint Infection
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Principal Investigator, Eugénie MABRUT, clinical research assistant, Hospices Civils de Lyon
Other Study IDs: 18-326
Record Dates: First submitted 2019-02-20; First posted 2019-02-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Bone and Joint Infection
Keywords: prosthetic joint infection; empirical antibiotherapy; acute kidney injury; vancomycin; cefepim; Piperacillin/tazobactam
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- empirical antibotherapy currently used: patients having had a vancomycin and piperacillin-tazobactam combination as empirical antibiotherapy
  Interventions: Other: empirical antibiotherapy
- another empirical antibotherapy: patients having had a vancomycin and cefepime combination as empirical antibiotherapy
  Interventions: Other: empirical antibiotherapy

INTERVENTIONS:
Other: empirical antibiotherapy — comparison of the outcome in the 2 groups having had 2 different empirical antibiotherapies

SUMMARY:
The empirical use of vancomycin in combination with a broad-spectrum beta-lactam is currently recommended after the initial surgery of prosthetic joint infection (PJI). However, the tolerability of such high-dose intravenous regimens is poorly known. T

DETAILED DESCRIPTION:
The empirical use of vancomycin in combination with a broad-spectrum beta-lactam is currently recommended after the initial surgery of prosthetic joint infection (PJI). However, the tolerability of such high-dose intravenous regimens is poorly known. The empirical antimicrobial therapy of PJI is associated with an important rate of adverse, linked with the use of the vancomycin and the piperacillin-tazobactam combination. Some studies suggest to use vancomycin-cefepime, which remains to be evaluated in PJI.

ELIGIBILITY:
Inclusion Criteria:

* patients having had a prosthetic joint infection and having had a postoperative empirical antibiotherapy with combination of vancomycine and piperacillin-tazobactam or vancomycine and cefepime

Exclusion Criteria:

* none

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients having had a prosthetic joint infection and having had a postoperative empirical antibiotherapy with combination of vancomycine and piperacillin-tazobactam or vancomycine and cefepime manage at the croix rousse hospital
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Rate of Treatment Failure | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption
  Treatment failure is defined by local clinical and/or microbiological relapse; and/or need for additional surgery; death of septic origin

SECONDARY OUTCOMES:
rate of adverse events | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption
  Description of adverses events leading to stop the empirical treatment
rate of bacteria responsible for infection | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption
  bacterial epidemiology

CONTACTS AND LOCATIONS:
Overall Officials: Florent Valour, Md,PhD, Study Director — HCL
Locations (1):
- Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided